CLINICAL TRIAL: NCT06680921
Title: A Randomized, Open-label, Phase III Study of SIM0270 Combined With Everolimus Versus Treatment of Physician's Choice in Patients With CDK4/6 Inhibitors Previously Treated , ER+/HER2- Locally Advanced or Metastatic Breast Cancer
Brief Title: A Study of SIM0270 Combined With Everolimus vs. Treatment of Physician's Choice in Patients With ER+/HER2- Advanced Breast Cancer (SIMRISE)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Collaborators: Nanjing Zaiming Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIM0270-301
Record Dates: First submitted 2024-11-05; First posted 2024-11-08 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Locally Advanced or Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Everolimus; exemestane; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): SIM0270 to be taken orally as a capsule in combination with Everolimus.
  Interventions: Drug: SIM0270; Drug: Everolimus (Afinitor®)
- Control group (Active Comparator): Investigator's choice of therapy of either:
  Fulvestrant alone (a solution for injection), or Everolimus in combination with exemestane, both a tablet to be taken orally.
  Interventions: Drug: Everolimus (Afinitor®); Drug: Exemestane tablets; Drug: Fulvestrant injection

INTERVENTIONS:
Drug: SIM0270 — Experimental
  Arms: Experimental group
Drug: Everolimus (Afinitor®) — Experimental and Active comparator
Drug: Exemestane tablets — Active Comparator
  Arms: Control group
Drug: Fulvestrant injection — Active Comparator
  Arms: Control group

SUMMARY:
This Phase III, randomized, open label, multicenter study will evaluate the efficacy and safety of SIM0270 combined with everolimus compared to physician's choice of treatment in subjects with ER+/HER2- locally advanced or metastatic breast cancer who have had previous treatment with CDK4/6 inhibitor.

ELIGIBILITY:
Inclusion criteria:

1. Subjects with histologically or cytologically confirmed ER+/HER2- locally advanced or metastatic breast cancer
2. Subjects must have at least one RECIST 1.1 measurable disease and /or at least 1 lytic or mixed (lytic + sclerotic) bone lesion
3. For women who are post menopausal must meet criteria as defined in the protocol.For women who are premenopausal or perimenopausal and for men: treatment with approved LHRH agonist therapy for screening period and the duration of study treatment
4. Have disease that has demonstrated progression on or after prior treatment:

   1. subjects had received 1 to 2 endocrine therapies in the locally advanced or metastatic setting with disease recurrence/disease progression while being treated with adjuvant endocrine therapy for ≥ 24 months and/or endocrine therapy in the locally advanced or metastatic setting, and derived a clinical benefit from therapy
   2. subjects had received ≤ 1 chemotherapy in the locally advanced or metastatic setting.
5. Eastern Cooperative Oncology Group Performance Status 0-1
6. Adequate organ function

exclusion criteria:

1. Prior treatment with a oral selective estrogen receptor degrader (SERD) or other investigational-ER-directed therapy, or any PI3K-AKI-mTOR inhibitors
2. Treatment with any investigational therapy within 28 days prior to study treatment.Treatment with moderate/strong CYP3A inhibitors or P-gP inhibitor within 14 days prior to first dose or moderate/strong CYP3A inducer within 28 days prior to first dose
3. Advanced, symptomatic, visceral spread that is at risk of life-threatening complications in the short term
4. Active or symptomatic CNS metastases, carcinomatous meningitis, or leptomeningeal disease
5. Active cardiac disease or history of cardiac dysfunction, as defined in the protocol
6. Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival(PFS) , as assessed by blinded independent review committee(BIRC) according to RECIST1.1 | 2 year
  PFS was defined as the time from the date of randomization to the first documented disease progression or death from any cause, whichever occurrs first.

SECONDARY OUTCOMES:
Progression free survival(PFS) , as assessed by investigator according to RECIST1.1 | 2 year
  PFS was defined as the time from the date of randomization to the first documented disease progression or death from any cause, whichever occurrs first.
Overall Survival (OS) | 3 year
  OS is the time from the date of randomization to death from any cause.
The incidence and severity of adverse events (AEs) and serious adverse events (SAEs) | 3 year
  Frequency and severity of Adverse Events or Serious Adverse Events as defined by CTCAE version 5.0
Blood concentrations | At five specified time points of the first 6 cycles (each cycle is 28 days)
  Blood concentrations of SIM0270 and everolimus
Objective Response Rate (ORR) by investigator | 2 year
  The objective response rate is defined as the percentage of subjects with a complete response or partial response.
Objective Response Rate (DOR) by investigator | 2 year
  The DoR is defined as the time from the date of first complete or partial response until the date of documented progression or death from any cause.
ORR by BIRC | 2 year
  The objective response rate is defined as the percentage of subjects with a complete response or partial response.
DOR by BIRC | 2 year
  The DoR is defined as the time from the date of first complete or partial response until the date of documented progression or death from any cause.
Clinical benefit rate(CBR) by investigator | 2 year
  The clinical benefit rate is defined as the percentage of subjects with a complete response or partial response or stable disease for ≥24 weeks.
CBR by BIRC | 2 year
  The clinical benefit rate is defined as the percentage of subjects with a complete response or partial response or stable disease for ≥24 weeks.
Time To Progression (TTP) by investigator | 2 year
  TTP is defined as the time from randomization until the date of first documented progression.
Time To Progression (TTP) by BIRC | 2 year
  TTP is defined as the time from randomization until the date of first documented progression.
Change from baseline in EQ-5D-5L scores | 2 year
  Change from baseline in EQ-5D-5L scores
Change from baseline in FACT-B scores | 2 year
  Change from baseline in FACT-B scores

CONTACTS AND LOCATIONS:
Locations (60):
- China (60):
  - The First Affiliated Hispital of Bengbu Medical University, Bengbu, Anhui
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - The First Affiliated Hispital of Anhui Medical University, Hefei, Anhui
  - Maanshan People's Hospital, Maanshan, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - The First Medical Center of PLA Ggeneral Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - The Second Affiliated Hospital of Fujian Medical University, Quanzhou, Fujian
  - Gansu Provincial Cancer Hospital, Lanzhou, Gansu
  - Guangdong Maternal and Child Health Hospital, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Zhongshan City People's Hospital, Zhongshan, Guangdong
  - Guangxi Medical University Cancer hospital, Nanning, Guangxi
  - First Hospital Of Qinhuangdao, Qinhuangdao, Hebei
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Anyang Tumor Hospital, Anyang, Henan
  - The First Affiliated Hospital of Henan University of Science & Technology, Luoyang, Henan
  - The Affiliated Cancer Hospital of Zhengzhou University and Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Wuhan Central Hospital, Wuhan, Hubei
  - Wuhan University Zhongnan Hospital, Wuhan, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - The First PEOPLE'S HOSPITAL OF CHANGDE CITY, Changde, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The Central Hospital of Yongzhou, Yongzhou, Hunan
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - The First Affiliated Hospital of JINZHOU Medical University, Jinzhou, Liaoning
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi
  - Baoji Central Hospital, Baoji, Shan'Xi
  - Binzhou Medical University Hospital, Binzhou, Shandong
  - Shandong First Medical University and Shandong Academy of Medical Sciences, Jinan, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - Linyi People'S Hostipal, Linyi, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Weifang People'S Hospital, Weifang, Shandong
  - Weihai Municipal Hospital, Weihai, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Ningbo Medical Center Lihuili Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided